CLINICAL TRIAL: NCT02922881
Title: Use of a Novel Diet (UC Diet) Targeting the Microbiota for Treatment of Mild to Moderate Active Pediatric Ulcerative Colitis: An Open Label Pilot Study
Brief Title: Microbiota-targeted Diet for Pediatric UC
Acronym: UCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Wolfson Medical Center (Other Government); IWK Health Centre (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-013075
Record Dates: First submitted 2016-06-13; First posted 2016-10-04 (Estimated); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ulcerative Colitis Diet (Experimental): Participants will receive a structured 12-week diet with a step down phase.
  Interventions: Other: Ulcerative Colitis Diet (UCD)

INTERVENTIONS:
Other: Ulcerative Colitis Diet (UCD) — The primary study intervention is a novel dietary intervention, the UC Diet. The UC Diet is a structured 12-week diet with a step down phase designed to remove products that allow harmful bacteria to thrive and add products that can change the bacteria in the gut to induce remission

SUMMARY:
Ulcerative colitis is a chronic inflammatory disease primarily involving the colon and has long been considered to be due to a dysregulated immune response targeting the colon, and involves unknown environmental factors. Currently, no effective therapy targets the microbiota or its interaction with the colonic epithelium. Diet has a significant impact on the composition of the microbiota; however, no dietary intervention to date has proven effective for induction of remission. The primary objective of this study is to determine whether the Ulcerative Colitis Diet (UCD) can induce remission or response in pediatric UC patients with active mild to moderate UC on a stable medication.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Established diagnosis of UC
* Age: 8-19 (inclusive)
* Mild to moderate active disease, 10<PUCAI<45
* Stable medication (IMM/5ASA) use or no medication use for the past 6 weeks.
* Participant has agreed to follow the UCD for 12 weeks

Exclusion Criteria:

* Any proven current infection such as positive stool culture, parasite or C. difficile within the past 4 weeks
* Antibiotic or corticosteroid use in the past 2 weeks
* Use of biologics in present or in the past
* PUCAI>45
* Acute severe UC in the previous 12 months
* Current extra intestinal manifestation of UC
* Primary Sclerosing Cholangitis (PSC) or liver disease
* Pregnancy
* Known food allergy to mandatory foods in the UCD

Ages: 8 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Clinical Remission | At 6 weeks following enrollment
  Remission defined by the Pediatric Ulcerative Colitis Activity Index (PUCAI)

SECONDARY OUTCOMES:
Dietary Compliance | Up to 12 weeks following enrollment
  Using modified Medication Adherence Rating Scale (MARS) questionnaire
Change in C-reactive protein (CRP) between baseline and week 12 | 12 weeks
Change in erythrocyte sedimentation rate (ESR) between baseline and week 12 | 12 weeks
Change in fecal calprotectin (FCP) between baseline and week 12 | 12 weeks
Microbial composition of the gastrointestinal tract | 12 weeks
  Change in the microbial composition of the stool and rectum from baseline to 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Albenberg, DO, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No